CLINICAL TRIAL: NCT06365398
Title: Safety and Efficacy of Low-dose Heparinization in Cerebral Angiography: a Randomized Controlled Study
Brief Title: Safety and Efficacy of Low-dose hEparinization in Cerebral Angiography sTudy
Acronym: SELECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SELECT; XWHL-2018010 (Other Grant/Funding Number: Xuanwu Hospital, Capital Medical University)
Record Dates: First submitted 2024-03-26; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2018-03

CONDITIONS: Cerebral Angiography; Heparinization
Keywords: cerebral angiography; heparin; Nursing; Ischemic Stroke; Safety; Efficacy
MeSH Terms: conditions — Ischemic Stroke | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: All patients enrolled are randomly divided into three groups according to the random number principle, which includes conventional systemic heparinization group, micro-dose systemic heparinization, and heparin-free angiography. It is carried out with a 1:1:1 ratio and variable block sizes.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular-dose group (Active Comparator): 3000~5000 Units of normal heparin was injected via the sheath tube in the systemic heparinization (Regular-dose) group. Half a dose of normal heparin is added after the imaging session has lasted more than half an hour.
  Interventions: Drug: Heparin
- Micro-dose group (Experimental): Micro-dose group is performed with two bags of 500 milliliter(ml) saline with 2500 Units of heparin were used to make a 5000 Units per liter heparin saline, which was used to infuse anticoagulation.
  Interventions: Drug: Heparin Sodium Injection
- heparinization group (Experimental): No heparinization is performed with no additional heparin is administered by a sheath or arterial route in the third group.
  Interventions: Other: No heparinization

INTERVENTIONS:
Drug: Heparin — As soon as the sheath was inserted, three different doses of heparin were administered according to the patients group assignment. In the conventional systemic heparinization (Regular-dose) group (The drug is Heparin Sodium Injection 2ml:12500 Units per bottle), systemic heparin was administered by intravenous injection at a dose of 83 Units/Kg. Patients in both the regular dose (83 units/kg) and low dose (42 units/kg) groups were given heparin intravenously once before the procedure of cerebral angiography, and no further heparin infusion was given during the angiography procedure. If the duration of the imaging procedure exceeded 1 hour, an additional 1/2 amount of the first dose of heparin was given.
  Other Names: Regular-dose heparinization
  Arms: Regular-dose group
Drug: Heparin Sodium Injection — In the micro-dose systemic heparinization (Micro-dose) group (the drug is Heparin Sodium Injection 2ml:12500 Units per bottle), systemic heparin was administered by intravenous injection at a dose of 42 Units/Kg. Patients in both the regular dose (83 units/kg) and low dose (42 units/kg) groups were given heparin intravenously once before the procedure of cerebral angiography, and no further heparin infusion was given during the angiography procedure. If the duration of the imaging procedure exceeded 1 hour, an additional 1/2 amount of the first dose of heparin was given.
  Other Names: Micro-dose heparinization
  Arms: Micro-dose group
Other: No heparinization — No additional heparin was administered via the sheath or arterial route in the no heparinization group.
  Arms: heparinization group

SUMMARY:
Purpose: Systemic heparinization is a widely used technique on digital subtraction angiography (DSA). Heparin, however, is associated with a variety of complications, including hemorrhage, thrombocytopenia, and hematomas. This study aimed to investigate the safety and efficacy of micro-dose systemic heparinization or no heparinization on cerebral angiography for cerebrovascular diseases.

Methods: A prospective, single-blind, randomized controlled study on patients who experienced transient ischemic attacks (TIAs) or acute ischemic strokes and underwent DSA is performed. Participants are randomized into three groups: regular-dose systemic heparinization, micro-dose systemic heparinization, and no heparinization. Information on patient demographics, laboratory tests, perioperative complications, and back pain scores is collected. Safety endpoints are defined as cerebral ischemic events and local complications of puncture site. Efficacy endpoints were defined as the recovery of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-65 years;
2. suspected cerebrovascular disease, including vascular lesions of the carotid, middle cerebral, anterior cerebral, vertebral, basilar, and posterior cerebral arteries;
3. Activity of daily living (ADL) score between 85~100;
4. normal coagulation function and no prior anticoagulant therapy before DSA;
5. fully informed consent to participate in the study.

Exclusion Criteria:

1. iodine allergy;
2. hepatic and/or renal insufficiency;
3. severe hypertension with poor blood pressure control;
4. hemorrhagic diseases;
5. hyperlipidemia;
6. poor glycemic control in diabetes;
7. pregnancy;
8. atrial fibrillation;
9. undergoing interventional treatment simultaneously.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
postoperative cerebral infarction | Perioperative period
  The safety endpoints of the study were postoperative cerebral infarction on imaging, and local complications such as bleeding at the puncture site, subcutaneous hematoma, and pseudoaneurysm diagnosed by computed tomography angiography (CTA). All patients underwent magnetic resonance imaging within 48 hours after cerebral angiography to check for new ischemic infarction. Postoperative ischemia was characterized as the abrupt appearance of novel neurological deficits, including hemiplegia, hemianopia, aphasia, dysphagia, sensory impairment, or confusion, persisting for more than 24 hours, accompanied with the presence of newly detected cerebral infarction using diffusion-weighted magnetic resonance imaging or computed tomography.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) for back pain | 24 hours after intervention
  Numerical Rating Scale (NRS) for back pain is assessed by investigators after intervention
the incidence of paralysis of surgical limb | 24 hours after intervention
  the incidence of paralysis is assessed after intervention
the incidence of pain of surgical limb | 24 hours after intervention
  the incidence of pain of surgical limb is assessed after intervention
the incidence of postoperative urethral catheterization | 24 hours after intervention
  the incidence of postoperative urethral catheterization is assessed after intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University., Beijing

REFERENCES:
- [Derived] Wang Z, Luo J, Qin Q, Tang H, Yao H, Wang T, Feng F, Li W, Sun M, Jiao L. Safety and efficacy of low dose or no heparinization in cerebral angiography: A randomized controlled study (SELECT trial). Brain Circ. 2024 Sep 13;11(4):301-308. doi: 10.4103/bc.bc_41_24. eCollection 2025 Oct-Dec. PMID 41531874